CLINICAL TRIAL: NCT02299700
Title: A Study to Preliminarily Assess the Janssen Autism Knowledge Engine in Children and Adults With Autism Spectrum Disorder
Brief Title: Study to Evaluate the Janssen Autism Knowledge Engine in Children and Adults With Autism Spectrum Disorder
Acronym: Mentis
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR104919; ASD-001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-09-29; First posted 2014-11-24 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Janssen Autism Knowledge Engine; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Autism Spectrum Disorder (ASD) Participants (6-9 years): Participants with ASD aged 6 to 9 years will be observed for the usability of the Janssen Autism Knowledge Engine (JAKE) personal healthcare record (pHR) and biosensors in stage 1 and stage 2 (at laboratory sites).
  Interventions: Other: No Intervention
- ASD Participants (13-17 years): Participants with ASD aged 13 to 17 years will be observed for the usability of the JAKE pHR and biosensors in stage 1 and stage 2 (at laboratory sites).
  Interventions: Other: No Intervention
- ASD Participants (3 or greater than 3 years): Participants with ASD aged 3 or greater than 3 years will be observed for the usability of the JAKE pHR and biosensors in stage 2 (at clinical sites).
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — The usability of the Janssen Autism Knowledge Engine (JAKE) as a system to monitor clinical outcomes in Autism Spectrum Disorder (ASD) will be observed.

SUMMARY:
The purpose of this study is to assess the usability of the Janssen Autism Knowledge Engine (JAKE) as a system to monitor clinical outcomes in autism spectrum disorder (ASD) (severe abnormalities in the development of many basic psychological functions that are not normal for any stage in development. These abnormalities are manifested in sustained social impairment, speech abnormalities, and peculiar motor movements).

DETAILED DESCRIPTION:
This is an observational (study in which participants identified as belonging to study groups are assessed for biomedical or health outcomes) and prospective (study following participants forward in time) study to determine JAKE in children and adults with ASD. The study will be conducted in 2 stages and each stage consists of 2 parts: Screening Phase (14 days), data collection Phase (Stage 1: 1 week and Stage 2: 4 weeks) and, stage 2 has follow-up Phase (up to 4 weeks post-data collection). The maximum study duration for each participant will not exceed 1 week for stage 1 and 8 weeks for stage 2. Primarily, the usability of JAKE as a system to monitor clinical outcomes in ASD will be assessed. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants can receive behavioral and/or pharmacologic treatments for Autism Spectrum Disorder (ASD) and comorbid disorders during the course of the study
* Parents or legally acceptable representatives must speak and understand English
* Participants must live with a parent or primary caregiver or, if not, they must either (A) spend at least 3 hours a day for at least 4 days each week or, (B) spend at least 3 weekends a month with a parent or primary caregiver
* Parents or legally acceptable representatives must possess (A) a portable electronic device capable of running the Janssen Autism Knowledge Engine (JAKE) application and connecting to the internet, and (B) a laptop or desktop computer connected to the internet
* In the opinion of the Investigator, participant and parents must be capable of completing all procedures and tasks of the study
* Diagnosis of ASD made or confirmed by the Investigator according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) criteria using a DSM V checklist and at least a 'mild' rating on the Child Autism Rating Scale 2 (CARS-2)

Exclusion Criteria:

* Lab sites only: Measured composite score on the Vineland Adaptive Behavior Scales (VABS) of less than 60
* History of or current significant medical illness that the Investigator considers should exclude the participant
* Psychological and/or emotional problems which would render the informed consent invalid or limit the ability of the participant to comply with the study requirements
* Any condition that in the opinion of the Investigator would complicate or compromise the study, or the wellbeing of the participant; for example, visual problems that would impede eye tracking or viewing the stimuli or hearing problems that would impede hearing auditory stimuli
* Employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and Adult participants with history of Autism Spectrum Disorder will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2015-04-24 (Actual)

PRIMARY OUTCOMES:
Stage 1: Usability of the Janssen Autism Knowledge Engine (JAKE) in Measuring Clinical Symptoms of Autism Spectrum Disorder (ASD) | Week 1
  The JAKE personal healthcare record (pHR) encompasses various modules for use by clinicians, caregivers, participants and the sponsor. The JAKE is accessible both through a web interface for computers and applications for mobile devices. The modules are medical/developmental history, symptom tracker, journal/ASD events, treatment tracker, dashboard, healthvault, research data warehouse and workbench. Results of several parent and clinician questionnaires will be compared with the findings of the mentis symptom tracker and biosensors. An exit survey will assess overall usability of the system.
Stage 2: Usability of the Janssen Autism Knowledge Engine (JAKE) in Measuring Clinical Symptoms of ASD | Week 4
  The JAKE personal healthcare record (pHR) encompasses various modules for use by clinicians, caregivers, participants and the sponsor. The JAKE is accessible both through a web interface for computers and applications for mobile devices. The modules are Medical/Developmental History, Symptom Tracker, Journal/ASD events, Treatment Tracker, Dashboard, HealthVault, Research Data Warehouse and Workbench. Results of several parent and clinician questionnaires will be compared with the findings of the mentis symptom tracker and biosensors. An exit survey will assess overall usability of the system.

SECONDARY OUTCOMES:
Utility of JAKE Symptom Tracker in Measuring Clinical Symptoms of ASD | Baseline and Week 1 in Stage 1, and Baseline and Week 4 in Stage 2
  The JAKE Symptom Tracker is a series of 97 questions related to the core and associated symptoms of ASD. Questions are answered on two 4-point scales, either frequency and intensity, frequency and context, or quality and context.
Correlation Between Key Biosensors and ASD Symptoms | Baseline and Week 1 in Stage 1, and Baseline and Week 4 in Stage 2
  The utility of the biosensors will be determined by measuring the associations between the biosensors and the ASD symptoms (response to tasks and stimuli in lab, the symptom tracker, and the event tracker).
Ease of use and Utility of JAKE for use in Prospective Clinical Trials | Baseline and Week 1 in Stage 1, and Baseline and Week 4 in Stage 2
  The JAKE personal healthcare record (pHR) encompasses various modules for use by clinicians, caregivers, participants and the sponsor. The JAKE is accessible both through a web interface for computers and applications for mobile devices. The modules are Medical/Developmental History, Symptom Tracker, Journal/ASD events, Treatment Tracker, Dashboard, HealthVault, Research Data Warehouse and Workbench.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 1 in Stage 1, and Up to Week 8 in Stage 2
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - Boston, Massachusetts
  - Toms River, New Jersey
  - Durham, North Carolina

REFERENCES:
- [Derived] Chatterjee M, Manyakov NV, Bangerter A, Kaliukhovich DA, Jagannatha S, Ness S, Pandina G. Learning Scan Paths of Eye Movement in Autism Spectrum Disorder. Stud Health Technol Inform. 2020 Jun 16;270:287-291. doi: 10.3233/SHTI200168. PMID 32570392
- [Derived] Bangerter A, Chatterjee M, Manfredonia J, Manyakov NV, Ness S, Boice MA, Skalkin A, Goodwin MS, Dawson G, Hendren R, Leventhal B, Shic F, Pandina G. Automated recognition of spontaneous facial expression in individuals with autism spectrum disorder: parsing response variability. Mol Autism. 2020 May 11;11(1):31. doi: 10.1186/s13229-020-00327-4. PMID 32393350
- [Derived] Bangerter A, Ness S, Lewin D, Aman MG, Esbensen AJ, Goodwin MS, Dawson G, Hendren R, Leventhal B, Shic F, Opler M, Ho KF, Pandina G. Clinical Validation of the Autism Behavior Inventory: Caregiver-Rated Assessment of Core and Associated Symptoms of Autism Spectrum Disorder. J Autism Dev Disord. 2020 Jun;50(6):2090-2101. doi: 10.1007/s10803-019-03965-7. PMID 30888551
- [Derived] Manfredonia J, Bangerter A, Manyakov NV, Ness S, Lewin D, Skalkin A, Boice M, Goodwin MS, Dawson G, Hendren R, Leventhal B, Shic F, Pandina G. Automatic Recognition of Posed Facial Expression of Emotion in Individuals with Autism Spectrum Disorder. J Autism Dev Disord. 2019 Jan;49(1):279-293. doi: 10.1007/s10803-018-3757-9. PMID 30298462
- [Derived] Manyakov NV, Bangerter A, Chatterjee M, Mason L, Ness S, Lewin D, Skalkin A, Boice M, Goodwin MS, Dawson G, Hendren R, Leventhal B, Shic F, Pandina G. Visual Exploration in Autism Spectrum Disorder: Exploring Age Differences and Dynamic Features Using Recurrence Quantification Analysis. Autism Res. 2018 Nov;11(11):1554-1566. doi: 10.1002/aur.2021. Epub 2018 Oct 1. PMID 30273450
- [Derived] Ness SL, Manyakov NV, Bangerter A, Lewin D, Jagannatha S, Boice M, Skalkin A, Dawson G, Janvier YM, Goodwin MS, Hendren R, Leventhal B, Shic F, Cioccia W, Pandina G. JAKE(R) Multimodal Data Capture System: Insights from an Observational Study of Autism Spectrum Disorder. Front Neurosci. 2017 Sep 26;11:517. doi: 10.3389/fnins.2017.00517. eCollection 2017. PMID 29018317